CLINICAL TRIAL: NCT03464188
Title: An Upstream Palliative Care Intervention for Rural Family Caregivers
Brief Title: An Upstream Palliative Care Intervention for Rural and African-American Advanced Cancer Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, James N Dionne-Odom, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: K99NR015903 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-13 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cancer, Metastatic; Family Members
Keywords: early palliative care; family caregiver; rural; African-American; telehealth
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care family caregiver participants will be informed of the UAB Comprehensive Cancer Center Patient and Family Resources webpage.
- Project Cornerstone (Experimental): The intervention is lay navigator-led with regular supervision by a specialist palliative care clinician. Regular caregiver distress thermometer screening and problem support and self-care coaching. Caregivers receive a Project Cornerstone Family Supporting Family (FSF) Binder that organizes intervention materials and contains educational information pertaining to the 6 base coaching sessions.
  Interventions: Behavioral: Project Cornerstone

INTERVENTIONS:
Behavioral: Project Cornerstone — Project Cornerstone basic elements are:
  1. The intervention is lay navigator-led with regular supervision by a specialist palliative care clinician;
  2. 6 base telephone/in-person sessions: Sessions cover specific topics (every 1-2 weeks, 20-60 minutes/session; by phone or in-person), followed by monthly follow-up and additional coaching sessions as needed;
  3. Regular caregiver distress thermometer screening and problem support and self-care coaching.
  4. Caregivers receive a Project Cornerstone Family Supporting Family (FSF) Binder that organizes intervention materials and contains educational information pertaining to the 6 base coaching sessions. Project Cornerstone begins within 60 days of a care recipient being diagnosed with advanced cancer and ends 1 year after care recipient death.
  Arms: Project Cornerstone

SUMMARY:
The burden placed on advanced cancer family caregivers (FCGs) and the toll on their mental and physical health have never been greater and is particularly pernicious for underserved groups in the Southeastern U.S., including rural-dwellers and African-Americans, for whom interventions have not been specifically developed and tested. The purpose of this K99/R00 is provide the awardee with the knowledge and training necessary to become a leading independent clinical investigator in developing and testing telehealth palliative care interventions for family caregivers (FCGs) of underserved persons with advanced cancer. The research specific aim during the K99 phase was to develop and tailor the content, format and delivery of a telehealth intervention for FCGs of persons with advanced cancer in the rural South. To meet this aim, qualitative semi-structured interviews were conducted with 26 lay healthcare navigators, 20 FCGs, and 18 patients with advanced cancer to elicit feedback on a FCG intervention outline based on published evidence-based interventions. After thematic analysis, major findings included that the intervention should: have topical content that is flexible and based on continuous assessment; include at least some face-to-face contact; cautiously consider internet-based technologies because internet access in rural areas is poor; and potentially have navigators lead the intervention with appropriate oversight and additional training. K99 study findings have been used to adapt and develop a potentially scalable FCG intervention in the Southern U.S. population (Project Cornerstone). The K99 study phase in combination with accomplishing the training objectives has successfully catalyzed the awardee's transition from a Postdoctoral Fellow to a Tenure-Track Assistant Professor at the University of Alabama at Birmingham School of Nursing. The overall goal during the R00 phase will be to conduct a small-scale pilot RCT of Cornerstone with 70 FCGs of rural-dwelling and/or African-American patients with advanced cancer to assess acceptability, feasibility, and potential efficacy. The research specific aims during the R00 phase are to: evaluate the acceptability of Cornerstone and the feasibility of enrolling and retaining 70 participants into a RCT of the FCG intervention for 24 weeks (Aim 1) and evaluate the potential efficacy of Cornerstone in improving caregiver (Aim 2) and care recipient (Aim 3) outcomes compared to usual care (quality of life and distress [anxiety/depressive symptoms]). The results will directly support an R-01 application to conduct an efficacy RCT of an early, telehealth PC intervention for Southern FCGs of underserved persons with advanced cancer.

DETAILED DESCRIPTION:
Enrollment goal was increased from 60 to 70 participants due to attrition.

ELIGIBILITY:
FAMILY CAREGIVERS

Inclusion Criteria:

1. ≥18 years of age;
2. Self-endorsing or identified by the patient as "a relative, friend, or partner that has a close relationship with you and who assists you with your medical care and who may or may not live in the same residence as you and who is not paid for their help";
3. Either caring for a patient: a) residing in a rural zip code (as classified by the U.S. Census' Rural-Urban Commuting Area [RUCA] system as small rural, large rural, and isolated [hereafter referred to as "rural"]) or b) who is African-American/Black;
4. Caring for a patient with advanced-stage cancer (see definition under Patient Inclusion criteria below); and
5. Caregivers will need NOT need to have an agreeable patient willing to participate in the study (for data collection only).
6. English-speaking and able to complete baseline measures.

Exclusion Criteria:

1) Self-reported severe mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse

PATIENTS

Inclusion Criteria:

1. ≥18 years of age;
2. Diagnosed within past 60 days of initial screening with an advanced cancer, defined as metastatic stage III/IV solid-tumor cancers of the lung, breast, gynecologic, head and neck, gastrointestinal, genitourinary cancer, and melanoma; and
3. Either: a) resides in a rural zip code or b) is African-American/Black.

Exclusion Criteria:

1) Medical record documentation of active severe mental illness (i.e., schizophrenia, bipolar disorder, or major depressive disorder), dementia, active suicidal ideation, uncorrected hearing loss, or active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of retaining 70 family caregiver-patient dyads | From date of enrollment to 24 weeks
  Proportion of participants completing study-related assessments from enrollment to 24 weeks
Feasibility of intervention completion | From date of enrollment to 24 weeks
  Proportion of participants completing core coaching sessions from enrollment to 24 weeks

SECONDARY OUTCOMES:
Family Caregiver Quality of Life | Baseline, week 8, and week 24
  The Caregiver Quality of Life Index- Cancer (CQOLC) scale is a 35-item cancer-specific instrument that assesses the carer of a cancer patient's quality of life, that is, some of the physical, social, emotional, and financial aspects of well-being, and functioning.
Family Caregiver Mood (Anxiety/Depressive Symptoms) | Baseline, week 8, and week 24
  This Hospital Anxiety and Depression Scale (HADS) is a 14-item scale, containing 7 items each for symptoms of depression and anxiety over the past 7 days. Subscale scores range from 0-21 with scores ≥8 indicating abnormally high symptoms.
Patient Quality of Life | Baseline, week 8, and week 24
  The Functional Assessment of Chronic Illness Therapy-Palliative Care (FACIT-Pal) is a 46-item scale, composed of physical, emotional, social, and functional well-being and additional concern subscales. Scores range from 0 to 184, where a higher score represents higher quality of life.
Patient Mood (Anxiety/Depressive Symptoms) | Baseline, week 8, and week 24
  This Hospital Anxiety and Depression Scale (HADS) is a 14-item scale, containing 7 items each for symptoms of depression and anxiety over the past 7 days. Subscale scores range from 0-21 with scores ≥8 indicating abnormally high symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James N Dionne-Odom, PhD, RN, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dionne-Odom JN, Azuero A, Taylor RA, Dosse C, Bechthold AC, Currie E, Reed RD, Harrell ER, Engler S, Ejem DB, Ivankova NV, Martin MY, Rocque GB, Williams GR, Bakitas MA. A lay navigator-led, early palliative care intervention for African American and rural family caregivers of individuals with advanced cancer (Project Cornerstone): Results of a pilot randomized trial. Cancer. 2022 Mar 15;128(6):1321-1330. doi: 10.1002/cncr.34044. Epub 2021 Dec 7. PMID 34874061